CLINICAL TRIAL: NCT04976738
Title: A Dose-ranging Study to Examine the Pharmacokinetics, Safety, Tolerability and Efficacy of Cybis™ 10:25 THC:CBD Oil in Adults With Chronic Back/Neck Pain
Brief Title: A Study of Cybis™ 10:25 THC:CBD Oil in Adults With Chronic Back/Neck Pain
Acronym: CYDEPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cymra Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYM-001-21
Record Dates: First submitted 2021-06-30; First posted 2021-07-26 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain; Neck Pain; Back Pain; Pain; Pain, Chronic; Pain, Back; Pain, Neck; CBD; THC
Keywords: medical cannabis; THC; CBD; chronic pain; neck pain; back pain; pain; dose-ranging; dose-finding
MeSH Terms: conditions — Chronic Pain; Neck Pain; Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm: Cybis™ 10:25 THC:CBD oil (Experimental): Cybis™ 10:25 THC:CBD oil administered oromucosally at doses varying from 0.5 mL once daily to 1.5 mL twice daily. Total duration of dosing is 28 days.
  Interventions: Drug: Cybis™ 10:25 THC:CBD oil

INTERVENTIONS:
Drug: Cybis™ 10:25 THC:CBD oil — Cybis™ 10:25 containing 10 mg/mL of D9-THC and 25 mg/mL of CBD, formulated in medium chain triglycerides (MCT)

SUMMARY:
This is a non-randomised, single arm, open-label study of medical cannabis, Cybis™ 10:25, in participants with chronic back or neck pain in which participants receive escalating doses of Cybis™ 10:25.

DETAILED DESCRIPTION:
This is a non-randomised, single arm, open-label study of Cybis™ 10:25 in participants with chronic back or neck pain in which participants receive escalating doses of Cybis™ 10:25.

The purpose of the study is to demonstrate the safety and tolerability of Cybis™ 10:25 in participants with moderate to severe chronic back or neck pain that is unresponsive to over-the-counter non-opioid analgesics.

Participants will undergo a screening visit, then seven clinic visits (Day 1, 2, 8, 15, 22, 29, and 35). Cybis™ 10:25 will be administered oromucosally at doses varying from 0.5 mL once daily to 1.5 mL twice daily. Total duration of dosing is 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years and less than 75 years of age on the date of the Screening Visit;
2. Have back and or neck pain of at least three months duration;
3. Have an average back or neck pain score of between 5 and 9 on a 10-point visual analogue pain scale;
4. Have failed to achieve self-reported satisfactory pain relief using over-the-counter paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs);
5. Are willing to cease all current pain medications 14 days prior to commencing Cybis™ 10:25, and for the duration of the study (except as allowed under rescue medication); Note: Pain medication may include opioids (including but not limited to paracetamol+codeine combinations, codeine, tramadol, tapentadol, buprenorphine), NSAIDs and other co-analgesic medications (such as anti-epileptics, antidepressants, clonidine) and/or any other pain medications.
6. Agree to cease any dietary or herbal supplements (e.g. St John's Wort) fourteen days prior to commencing Cybis™ 10:25, and for the duration of the study;
7. Are willing to cease driving a car or operating heavy machinery from the day of first dosing to seven days after administration of the last dose of Cybis™ 10:25;
8. Agree to use contraception throughout the study, and for one month after the last dose of Cybis™ 10:25 is administered (if reproductive age female) or three months after the last dose of Cybis™ 10:25 is administered (if male); Note: women of childbearing potential must have a negative serum or urine pregnancy test prior to entry into the study. For women, adequate contraception is a double barrier method for the duration of the study and for 30 days post the last study dose. For men, barrier contraception is required for the duration of the study and for 3 months after the last study dose.
9. Agree to adhere to the study protocol; and
10. Are willing and able to provide written informed consent.

Exclusion Criteria:

1. Are pregnant or breastfeeding;
2. Currently using marijuana or other medicinal cannabis products; Use of medical cannabis products > 6 months prior to Screening is acceptable;
3. History of cannabis use disorder (score of 8 or higher on The Cannabis Use Disorder Identification Test - Revised (CUDIT-R);
4. Current or previous allergies or allergic responses to any of the components of the study treatment (e.g., THC, CBD, MCT);
5. Current or previous allergies or allergic responses to any of the components of the rescue medication (e.g. paracetamol, ibuprofen, aspirin, other NSAIDs);
6. Significant cardiac disease (e.g. poorly controlled hypertension, symptomatic ischaemic heart disease, symptomatic heart failure);
7. Chronic liver disease with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper level or normal limits;
8. Chronic renal impairment with eGFR <30mL/min;
9. Taking sildenafil or other PDE5 inhibitors;
10. Being treated with known inducers/inhibitors of CYP3A4, in particular clarithromycin, rifampicin, azole antifungals, antiretroviral agents, anticonvulsants (phenytoin, carbamazepine), SSRI within 30 days of study commencement; Use of such enzyme-altering agents is prohibited throughout the study.
11. Have a major psychiatric disorder (e.g. schizophrenia, psychosis, bipolar disorder, but not anxiety or depression), by history or examination;
12. Are currently using any illicit drug (including, but not limited to, amphetamines, cocaine);
13. Have a history of other substance abuse disorder (as defined by DSM-5);
14. Have active substance abuse disorder (alcohol, illicit drugs);
15. Other clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, or vital signs, which in the opinion of the Investigator, may put the participant at risk of adverse events;
16. Other chronic disease (other than chronic pain) that in the opinion of the Investigator may impact the safety, efficacy and/or pharmacokinetics of the study drug;
17. Are currently participating in, or have participated (in the last 30 days) in a drug or device clinical trial;
18. Currently using opioids (including but not limited to paracetamol+codeine combinations, codeine, tramadol, tapentadol, buprenorphine) and not willing to cease opioids for the duration of the study;
19. COVID-19 vaccination within two (2) weeks of study assessments:

    1. Study assessments should not commence until two (2) weeks after a COVID-19 vaccination dose (first, second or booster dose)
    2. Subsequent COVID-19 vaccination doses (first, second or booster dose) should not be administered until 7 days after Day 35 study assessments have been completed.
20. Back and/or neck surgery within three (3) months of Screening; or
21. Have history of metastatic cancer or are currently receiving treatment for cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Number (and percentage) of participants with one or more adverse event | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants with one or more adverse event of special interest | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants with one or more serious adverse events | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Adverse events, adverse events of special interest, serious adverse events will be summarised descriptively with the number of participants experiencing the event and the percentages of participants experiencing the event. | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants with changes in vital signs | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants with clinically relevant changes in physical examination | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants with clinically relevant changes in clinical chemistry | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants who drop-out | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.
Number (and percentage) of participants who withdraw due to adverse events | Safety and tolerability will be assessed throughout the trial. Up to 35 days.
  To assess the safety and tolerability of Cybis™ 10:25 at low (0.5 mL qd), medium-low (0.5 mL bd), medium (1.0 mL bd) and high (1.5 mL bd) doses.

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. Peak plasma concentration (Cmax) of THC in plasma. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The concentration at peak (Cmax) will be calculated for THC. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. Time to maximum concentration (tmax) of THC in plasma. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The time to reach peak (tmax) will be calculated for THC. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. Area under the concentration/time curve (AUC) will be calculated for THC. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The area under the concentration/time curve (AUC) will be calculated for THC. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The elimination half-life (t1/2) will be calculated for THC. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The elimination half-life (t1/2) will be calculated for THC. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. Peak plasma concentration (Cmax) of CBD in plasma. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The concentration at peak (Cmax) will be calculated for CBD. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. Time to maximum concentration (tmax) of CBD in plasma. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The Time to maximum concentration (tmax) will be calculated for CBD. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The area under the concentration/time curve (AUC) will be calculated for CBD. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The area under the concentration/time curve (AUC) will be calculated for CBD. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The elimination half-life (t1/2) will be calculated for CBD. | Up to 29 days. Samples collected at baseline 0 (pre-dose), 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 9.0, 12.0, and 24.0 hours post dosing. Day 8, 15, 22 and 29 trough levels.
  To investigate the pharmacokinetics of Cybis™ 10:25 in participants with chronic back and neck pain following single and repeated doses. The elimination half-life (t1/2) will be calculated for CBD. Pharmacokinetic calculations will be conducted for each dose level individually.
To investigate the dose-response relationship between Cybis™ 10:25 and pain response, as measured by the change from baseline in Numerical Pain Rating Scale (NPRS) | Baseline (pre-dose), Day 1, 8, 15, 22, 29 and 35
  To investigate the dose-response relationship between Cybis™ 10:25 and pain response as measured by the change from baseline in Numerical Pain Rating Scale (NPRS).
  The NPRS is an 11-point scale between 0 (no pain) and 10 (worst pain ever possible). The minimum clinically significant change in NPRS is two points. The NPRS has been validated for use in participant with low back pain.
  Baseline pain levels are considered the NPRS at Day 1, irrespective of dose cohort. Change from baseline will be calculated as the pain level at the end of a dose cohort (Day 8 for 0.5 mL once daily; Day 15 for 0.5 mL bd; Day 22 for 1.0 mL bd; or Day 29 for 1.5 mL bd) minus the Day 1 value.
To investigate the dose-response relationship between Cybis™ 10:25 and pain response, as measured by the change from baseline in Brief Pain Inventory - Short Form. | Baseline (pre-dose), Day 1, 8, 15, 22, 29 and 35
  To investigate the dose-response relationship between Cybis™ 10:25 and pain response as measured by the change from baseline in Brief Pain Inventory - Short Form.
  The Brief Pain Inventory-Short Form is a questionnaire that assesses worst pain in the last 24 hours, least pain in the last 24 hours, average pain, and pain 'right now' along with the interference the pain causes on general activity, mood, walking ability, normal work, relations with others, sleep and enjoyment of life. It will be scored according to its scoring manual [24]. Scores will be summarised at baseline, Day 8, 15, 22, 29 and 35.
To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in Depression Anxiety Stress Scale. | Baseline (pre-dose), Day 1, 8, 15, 22, 29 and 35
  To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in Depression Anxiety Stress Scale.
  The Depression Anxiety Stress Scale (DASS) is a 21-item self-report instrument used to measure depression, anxiety and stress. The DASS will be scored according to its scoring manual. Participants will be categorised as having normal, mild, moderate, severe, or extremely severe symptoms. Lower scores indicate normal symptoms, whereas higher scores indicate severe symptoms.
  Changes from baseline in DASS subscale scores will be used to investigate the dose-response relationship.
To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in Medical Outcomes Sleep Survey. | Baseline (pre-dose), Day 1, 8, 15, 22, 29 and 35
  To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in Medical Outcomes Sleep Survey.
  The Medical Outcomes Sleep Scale is a 12-item scale that assesses sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. It will be scored according to its scoring manual.
  The change in MOS Sleep Problems Index will be used to investigate the dose-response relationship.
To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in Self-Assessment of Treatment (SAT-II) scale. | Baseline (pre-dose), Day 1, 8, 15, 22, 29 and 35
  To investigate the dose-response relationship between Cybis™ 10:25 and quality of life as measured by the change from baseline in in Self-Assessment of Treatment (SAT-II) scale.
  The Self-Assessment of Treatment is a 9-item scale that measures treatment satisfaction in the previous seven days. It assesses pain, self-care activities, daily activities, physical activities, emotional well-being, sleep and social functioning, all assessed on a 5-point Likert scale. It also captures how likely the respondent would be willing to receive the study treatment again, and how study treatment compares to other treatments. The SAT-II has been validated, and is considered an acceptable endpoint for pain studies. The change in Self-Assessment of Treatment score will be used to investigate the dose-response relationship.
To investigate rescue medication use in participants prescribed Cybis™ 10:25 (proportion of patients requiring rescue medication, the number of doses of rescue medication required, the time to rescue medication). | Day 1, 8, 15, 22, 29 and 35
  To investigate rescue medication use in participants prescribed Cybis™ 10:25 for chronic back and neck pain.
  The proportion of patients requiring rescue medication and the number of doses of rescue medication required will be analysed descriptively. The time to first dose of rescue medication will be calculated using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chye, Study Director — Cymra Life Sciences
Locations (2):
- Australia (2):
  - ACRN - Australian Clinical Research Network, Maroubra, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No